CLINICAL TRIAL: NCT02300467
Title: A Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of NOV120401 (CKD-516 Tablet) in Patients With Advanced Refractory Solid Tumors
Brief Title: NOV120401 (CKD-516 Tablet) for Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National OncoVenture (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV120401-101
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Advanced Refractory Solid Tumors
MeSH Terms: interventions — N-(4-(3-(1H-1,2,4-triazol-1-yl)-4-(3,4,5-trimethoxybenzoyl)phenyl)thiazol-2-yl)-2-amino-3-methylbutanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOV120401 (CKD-516 Tablet) (Experimental): 5 to 45 mg/day PO for 5 consecutive days and 2 days off
  Interventions: Drug: NOV120401

INTERVENTIONS:
Drug: NOV120401 — 5 to 45 mg/day PO for 5 consecutive days and 2 days off
  Other Names: CKD-516 Tablet

SUMMARY:
The purpose of this open-label, dose-escalation phase I trial is to evaluate the safety, tolerability and pharmacokinetic profiles and to assess the efficacy of NOV120401 (CKD-516 Tablet), a novel vascular disrupting agent, in patients with advanced refractory solid tumors.

DETAILED DESCRIPTION:
Vascular disrupting agents are expected to kill cancer cells located in core of tumor tissues by disrupting microvascular structure of tumor. To assess the safety and tolerability of NOV120401 (CKD-516 Tablet), patients with advanced refractory solid tumors will be enrolled in this study. Initial dose of NOV120401 (CKD-516 Tablet) is 5 mg/day, which will be escalated until at least 2 of 6 subjects show dose-limiting toxicities (DLTs). Pharmacokinetic profiles and efficacy by tumor response and vascular disrupting activities will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 19 years or older
2. Patients who failed existing anti-cancer therapies
3. ECOG performance status ≤ 2
4. Life expectancy of ≥ 12 weeks
5. Adequate hematological, hepatic and renal functions:
6. Patients who give written informed consent voluntarily

Exclusion Criteria:

1. Prior systemic chemo-, radiochemo-, radio-, immuno-, hormonal and/or biological therapy within 2 weeks before study participation (in case of nitrosoureas and/or mitomycin, within 6 weeks before study participation)
2. Patients who received major surgery within 4 weeks before study participation (in case of VATS and/or ONC surgery, within 2 weeks before study participation)
3. Symptomatic CNS metastases (patients with radiologically and neurologically stable metastases and being off corticosteroids for at least 4 weeks are able to participate in this trial.)
4. NYHA class III or IV heart failure, uncontrolled hypertension (SBP/DBP > 140/90 mm Hg), other clinically significant cardiovascular abnormalities at investigator's discretion (e.g., LVEF < 50%, clinically significant cardiac wall abnormalities or cardiac muscle damages)
5. Acute coronary syndrome (unstable angina or myocardial infarction) within 6 months
6. Uncontrolled arrhythmia
7. Significant cerebrovascular diseases including stroke within 6 months
8. Significant vascular diseases including aortic aneurysm requiring treatment or peripheral arterial diseases
9. Patients with known active hepatitis, HIV infection, or other uncontrolled infectious disease
10. Patients who cannot receive IP by mouth and have a history of clinically significant gastrointestinal disorders which can impede administration, transit or absorption of the IP
11. A history of severe drug hypersensitivity or hypersensitivity to analogs of the IP
12. Pregnancy or breast-feeding
13. Women of childbearing potential (WOCBP) or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 2 months after the end of treatment
14. Patients who received other investigational products or used other investigational devices within 3 weeks before participation
15. Patients who cannot participate in this trial by investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Safety and MTD/recommended phase 2 dose (RP2D) determination (Number of Participants with Adverse Events) | By 40 weeks after enrollment of the last subject
  Number of Participants with Adverse Events

SECONDARY OUTCOMES:
Pharmacokinetic profiles (Cmax, Tmax, AUClast, AUCinf, t1/2, CL, MRT, Ctrough) of CKD-516 and S516 (active metabolite of CKD-516) | 21 days
Tumor response | up to 36 weeks
Vascular disrupting activity measured by tubulin status (western blot from peripheral blood mononuclear cell) | 21 days
  western blot from peripheral blood mononuclear cell
Vascular disrupting activity measured by plasma factor (VEGF, G-CSF, GM-CSF, SDF-1) concentration from serum | 21 days
  concentration from serum

CONTACTS AND LOCATIONS:
Overall Officials: Jung Yong Kim, MD, Study Director — National OncoVenture (jyk1949@ncc.re.kr); Min Chae Kim, Pharmacist, Study Director — National OncoVenture (minchae@ncc.re.kr)
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea